CLINICAL TRIAL: NCT02281110
Title: A Prospective, Observational, Non-randomized European, Multi-center Registry Collecting Real Life Information for the Utilization of Instantaneous Wave Free Ratio in Assessing Coronary Stenosis Relevance in the Multi-vessel Disease Patients Population.
Brief Title: The REAL Registry for Utilization of iFR in Assessing Coronary Stenoses
Acronym: DEFINE REAL
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-CV-001
Record Dates: First submitted 2014-10-01; First posted 2014-11-03 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Disease
Keywords: Diagnostic coronary catheterization; Multi-vessel coronary disease; Percutaneous Coronary Intervention; Instantaneous wave free ratio; Fractional flow reserve
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- iFR/FFR assessment: Patients enrolled into this prospective registry will be derived from Stable Coronary Artery disease or Acute Coronary Syndrome (ACS) population undergoing cardiac catheterization. Patients with ACS may be evaluated by functional assessment in the non-culprit stenosis during the index PCI revascularization or in a staged procedure. The registry will enroll patients in whom physiological assessment (iFR/FFR) is particularly helpful in identifying haemodynamically significant stenosis: MVD patients defined by patients with lesions > 40% and <100% in 2 or more vessels.
  Interventions: Device: iFR/FFR

INTERVENTIONS:
Device: iFR/FFR — • The Volcano iFR®-FFR option, which is a measurement modality for the Volcano system that provides the capability to make FFR and instantaneous wave-Free Ratio™ (iFR®) measurements (CE-Marked). iFR® is a pressure-derived, hyperemia-free index for the assessment of coronary stenosis relevance. This option consists of an FFR-iFR® specific patient interface module (PIM-FFR) which can be connected to the Volcano system - VOLCANO s5 or s5i™ platform equipped with iFR® option. This PIM-FFR is compatible with all Volcano pressure measurement guide wires.
  Other Names: instant flow reserve/fractional flow reserve

SUMMARY:
The purpose of this registry is to collect real life information and to document the performance and user friendliness of iFR in daily diagnostic practice and treatment strategies for MVD patients undergoing cardiac catheterization.

DETAILED DESCRIPTION:
The REAL Registry will enroll a maximum of 3,000 patients in approximately 300 sites across multiple European and Middle East countries, where product has received CE approval and is marketed. An average of 10 cases with a maximum of 50 patients will be enrolled per participating site.

No follow-up will be performed. The REAL Registry will only collect data during diagnostic angiogram or PCI procedure, when performed.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 year of age
* Willing to participate and able to understand, read and sign the informed consent document before the planned procedure
* Eligible for coronary angiography and PCI
* Coronary artery disease with at least two or more visually assessed coronary stenoses (greater than 40% diameter stenosis) in native, major epicardial vessel or its branches by coronary angiogram with an indication of physiological assessment.

Exclusion Criteria:

* Inability to obtain a signed informed consent from potential patient.
* Any contraindication for functional assessment as per the instructions per use and determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibility includes adults undergoing coronary angiography and/or PCI
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hemodynamic severity (Percentage of stenosis properly classified by iFR®) | Day 1 (Post-Procedure)
  Percentage of stenosis properly classified by iFR® in terms of hemodynamic severity compare to FFR in MVD patients. Hemodynamic severity will be established with an FFR value <=0,80.

SECONDARY OUTCOMES:
changes in iFR® and FFR | Day 1 (Post-Procedure)
  Changes in iFR® and FFR pre angioplasty and post angioplasty in MVD patients.
Changes to decision strategy of revascularization | Day 1 (Post-Procedure)
  Percentage of MVD patients in whom the decision strategy of revascularization changed after iFR® compare to the decision based on diagnostic angiogram only.

CONTACTS AND LOCATIONS:
Locations (1):
- Volcano Europe BVBA/SPRL, Zaventem, Belgium